CLINICAL TRIAL: NCT05033457
Title: Comparative Study Between Unilateral Biportal Endoscopy Technique and Percutaneous Endoscopic Transforaminal Discectomy for the Treatment of Lumbar Spinal Canal Stenosis
Brief Title: Comparative Study Between UBE and PETD for the Treatment of Lumbar Spinal Canal Stenosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Shaanxi Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Rongcan Liu, Director, Shaanxi Provincial People's Hospital
Other Study IDs: sxsrmyyjzwc202101
Record Dates: First submitted 2021-08-09; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-01

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- unilateral biportal endoscopy technique group: Treatment of lumbar intervertebral disc herniation with unilateral biportal endoscopy technique in unilateral biportal endoscopy technique group
  Interventions: Procedure: unilateral biportal endoscopy technique or percutaneous endoscopic transforaminal discectomy
- percutaneous endoscopic transforaminal discectomy group: Treatment of lumbar intervertebral disc herniation with percutaneous endoscopic transforaminal discectomy in percutaneous endoscopic transforaminal discectomy group
  Interventions: Procedure: unilateral biportal endoscopy technique or percutaneous endoscopic transforaminal discectomy

INTERVENTIONS:
Procedure: unilateral biportal endoscopy technique or percutaneous endoscopic transforaminal discectomy — Treatment of lumbar intervertebral disc herniation with unilateral biportal endoscopy technique in unilateral biportal endoscopy technique group.Treatment of lumbar intervertebral disc herniation with percutaneous endoscopic transforaminal discectomy in percutaneous endoscopic transforaminal discectomy group.

SUMMARY:
OBJECTIVE Both unilateral biportal endoscopy technique(UBE) and percutaneous endoscopic transforaminal discectomy(PETD) are minimally invasive and effective surgical procedures for lumbar spinal stenosis.The object of this retrospective study was to compare the clinical and radiological outcomes between UBE and PETD.

METHODS In the period from July 2020 to December 2020, using UBE or PETD to treat lumbar canal stenosis.Patients were classified into two groups based on the surgery they had undergone. Preoperative and postoperative MR image was used to evaluate the removal rate of lumbar disc herniated material by two surgical methods. The two surgical methods are also compared and evaluated in terms of operation time, incision size, hospitalization time, etc.

DETAILED DESCRIPTION:
It was performed as a retrospective analysis of prospectively collected data on patients received spinal endoscopic decompression between July 2020 to December 2020 was conducted. All patients underwent lumbar MRI examination with the result of L5-S1 disc herniation，accompanied by claudication or lower extremity radiation pain and other nerve compression symptoms. The symptoms have not improved with conservative treatments including physical therapy, medication, and epidural injection procedures for a minimum of 12 weeks. Patients who hadprevious spine surgery, infection, trauma, tumors or spondylolisthesis were excluded. The surgery was performed by the same experienced spinal surgeon and the surgical patient were closely followed for 3 months after surgery.

The investigators performed two kinds of endoscopic lumbar discectomy：unilateral biportal endoscopy technique(UBE) and percutaneous endoscopic transforaminal discectomy(PETD).

ELIGIBILITY:
Inclusion Criteria:

- Single-segment lumbar disc herniation/lumbar spinal stenosis

Exclusion Criteria:

* Multi-segment lumbar disc herniation / lumbar spinal stenosis、Have received surgery、Hypertension、Diabetes

Inclusion Criteria:

Inclusion Criteria:

Single-segment lumbar disc herniation Symptoms of nerve compression

Exclusion Criteria:

foraminal and extraforaminal disc herniation multilevel disc herniation, spinal stenosis spondylolisthesis scoliosis prior lumbar surgery spinal infection spinal tumor a history of hip or knee arthritis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with lumbar spinal stenosis, with low back pain and neurological urgency.The patient cannot relieve symptoms after 3 months or more of conservative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional area of the preoperative lumbar intervertebral disc | preoperative
  The preoperative axial T2-weighted MRI slices of the patient can be used to measure the cross-sectional area of the intervertebral disc of the diseased segment.
Cross-sectional area of the preoperative spinal canal | preoperative
  The preoperative axial T2-weighted MRI slices of the patient can be used to measure the cross-sectional area of the spinal canal of the diseased segment.
Cross-sectional area of the postoperative lumbar intervertebral disc | 3 months after surgery
  The postoperative axial T2-weighted MRI slices of the patient can be used to measure the cross-sectional area of the intervertebral disc of the diseased segment.
preoperative ODI | preoperative
  According to the Oswestry Disability Index (ODI), evaluate the preoperative ODI of participants.
ODI on 3 months after operation | 3 months after surgery
  According to the Oswestry Disability Index (ODI), evaluate the ODI of participants on 3 months after operation.
ODI at the final follow-up | Final follow-up
  According to the Oswestry Disability Index (ODI), evaluate the ODI of participants at the final follow-up.
preoperative VAS back pain score | preoperative
  According to the visual analog scale (VAS) scoring standard, assess the preoperative VAS back pain score of participants.
preoperative VAS leg pain score | preoperative
  According to the visual analog scale (VAS) scoring standard, assess the preoperative VAS leg pain score of participants.
VAS back pain score on postoperative day 1 | 1 day after operation
  According to the visual analog scale (VAS) scoring standard, assess the VAS back pain score of participants on postoperative day 1.
VAS leg pain score on postoperative day 1 | 1 day after operation
  According to the visual analog scale (VAS) scoring standard, assess the VAS leg pain score of participants on postoperative day 1.
VAS back pain score on 3 months after operation | 3 months after operation
  According to the visual analog scale (VAS) scoring standard, assess the VAS back pain score of participants on 3 months after operation.
VAS leg pain score on 3 months after operation | 3 months after operation
  According to the visual analog scale (VAS) scoring standard, assess the VAS leg pain score of participants on 3 months after operation.
VAS back pain score at the final follow-up | Final follow-up
  According to the visual analog scale (VAS) scoring standard, assess the VAS back pain score of participants at the final follow-up.
VAS leg pain score at the final follow-up | Final follow-up
  According to the visual analog scale (VAS) scoring standard, assess the VAS leg pain score of participants at the final follow-up.

SECONDARY OUTCOMES:
operation time | intraoperative
  Collect the operation time of participants during the operation.
incision size | intraoperative
  Collect the incision size of participants during the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jingpeng Wei, Study Chair — Shanxi Medical University
Locations (1):
- Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided